CLINICAL TRIAL: NCT02340169
Title: An Open Label, Safety Study to Assess the Potential for Adrenal Suppression and Pharmacokinetics Following Maximal Use Treatment With Topicort® (Desoximetasone) Topical Spray, 0.25% in Pediatric Patients With Plaque Psoriasis.
Brief Title: Adrenal Suppression and Pharmacokinetics of Topicort® Spray, 0.25% in Pediatric Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSXS-1303
Record Dates: First submitted 2014-12-28; First posted 2015-01-16 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Desoximetasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topicort® Topical Spray, 0.25% (Experimental): Topicort® (desoximetasone) Topical Spray, 0.25%, twice a day for 28 days
  Interventions: Drug: Topicort® (desoximetasone) Topical Spray, 0.25%

INTERVENTIONS:
Drug: Topicort® (desoximetasone) Topical Spray, 0.25% — Topicort® (desoximetasone) Topical Spray, 0.25% applied to affected areas twice a day for 28 days
  Other Names: desoximetasone

SUMMARY:
The objective of this study is to evaluate the potential of Topicort® (desoximetasone) Topical Spray, 0.25% to suppress hypothalmic pituitary adrenal axis function. The secondary objectives are to evaluate the efficacy parameters, pharmacokinetics and adverse event profile.

DETAILED DESCRIPTION:
An open label, post marketing safety study to assess the potential of a TOPICORT® (desoximetasone) Topical Spray, 0.25% to suppress HPA axis function following twice daily dosing for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 7 years and older must have provided written assent accompanied by written informed consent from patient's representative
* Clinical diagnosis of stable plaque psoriasis with involvement of ≥ 10% body surface area (excluding face and scalp)
* Physicians Global Assessment score of 3 or 4 at baseline

Exclusion Criteria:

* Has other dermatological conditions that may interfere with clinical assessments
* Allergy or sensitivity to corticosteroids or any drug hypersensitivity or intolerance that would compromise patient safety or study results
* History of an adverse reaction to Cortrosyn™ or similar test reagents
* Chronic infectious disease, system or organ disorder or other medical condition that would place patient at undue risk by study participation

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient enrolled in the study 23 January 2015. The last patient completed the study 22 November 2019. The Patients were enrolled in 3 cohorts. Cohort 1, 12 to 17 years and 11 months, Cohort 2, 6 year to 11 and 11 Months and Cohort 3, 2 years to 5 years and 11 months. In total 129 subjects were enrolled across 7 Investigator sites.
Pre-assignment Details: Prior to the Protocol Amendment if a subject was found to have an abnormal adrenal function test after the baseline Cortisol Response test the subject was notified to discontinue the drug and follow up with the Investigator. After the protocol amendment a screening visit was added so that subjects with abnormal tests would not be randomized to study drug.
Period: Overall Study
Arm/Group | Topicort® Topical Spray, 0.25%
Started | 129
Cohort 1 12-17 Years of Age | 84
Cohort 2 6 to 11 Years of Age | 35
Cohort 3 2 to 5 Years of Age | 10
Completed | 106
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Topicort® Topical Spray, 0.25%
Number analyzed (Participants) | 129
Age, Customized [Count of Participants; unit: Participants]
  Cohort 1 - 12 to 17 years of age | 84
  Cohort 2- 6 to 11 years of age | 35
  Cohort 3 - 2 to 5 years of age | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Population: the participants were analyzed in three separate cohorts
  Participants
    Cohort 1 -12 to 17 years of age: number analyzed (Participants) | 84
    Cohort 1 -12 to 17 years of age: Female | 35
    Cohort 1 -12 to 17 years of age: Male | 49
    Cohort 2 - 6 to 11 years of age: number analyzed (Participants) | 35
    Cohort 2 - 6 to 11 years of age: Female | 23
    Cohort 2 - 6 to 11 years of age: Male | 12
    Cohort 3- 2 to 5 years of age: number analyzed (Participants) | 10
    Cohort 3- 2 to 5 years of age: Female | 4
    Cohort 3- 2 to 5 years of age: Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 126
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 102
  More than one race | 0
  Unknown or Not Reported | 26
Region of Enrollment [Number; unit: participants]
  United States | 76
  Panama | 27
  El Salvador | 26
Hypothalamic-Pituitary-Adrenal (HPA) Axis Function [Count of Participants; unit: Participants] — HPA axis suppression was measured in the 100 evaluable subjects. Population: HPA Axis suppression was measured in the 100 evaluable subjects.
  Participants
    Cohort 1 - 12 to 17 years of age: number analyzed (Participants) | 84
    Cohort 1 - 12 to 17 years of age | 60
    Cohort 2 - 6 to 11 years of age: number analyzed (Participants) | 35
    Cohort 2 - 6 to 11 years of age | 30
    Cohort 3 - 2 to 5 years of age: number analyzed (Participants) | 10
    Cohort 3 - 2 to 5 years of age | 10

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Hypothalmic Pituitary Adrenal Axis Function Suppression as Measured by Cortisol Response Test
Description: A patient will be considered to have potential HPA axis suppression if they meet at least one of the criteria:
  * their 30 minute post injection cortisol level is not at least 7 mcg/100 ml greater than the basal level (< basal + 7)
  * the post stimulation level is ≤ 18 mcg/100 ml
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: 12 to 17 Years of Age
- Cohort 2: 6 to 11 Years of age
- Cohort 3: 2 to 5 years of age
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 60 | 30 | 10
Participants | 21 | 13 | 2
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other; Adrenal suppression rates in the evaluable population were 35% (21 out of 60), 43.3% (13 out of 30) and 20% (2 out of 10) in Cohorts 1, 2 a nd 3, respectively

2. Secondary Outcome: Adverse Event
Description: The total number of subjects experiencing adverse events.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Topicort® Topical Spray, 0.25%
Number analyzed (Participants) | 129
Participants | 1

3. Secondary Outcome: Cpre-ss
Description: Concentration prior to dosing at steady state.
Time Frame: 28 Days
Population: PK sampling from was taken from a subset of patients in cohorts 1 and 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Topicort® Topical Spray, 0.25% - Cohort 1; Topicort® Topical Spray, 0.25% - Cohort 2: Topicort® (desoximetasone) Topical Spray, 0.25%, twice a day for 28 days
  Topicort® (desoximetasone) Topical Spray, 0.25%: Topicort® (desoximetasone) Topical Spray, 0.25% applied to affected areas twice a day for 28 days
Arm/Group | Topicort® Topical Spray, 0.25% - Cohort 1 | Topicort® Topical Spray, 0.25% - Cohort 2
Number analyzed (Participants) | 11 | 8
pg/mL | 527.64 (574.47) | 475.41 (215.66)

ADVERSE EVENTS:
Time Frame: For each subject Adverse Events were collected during their 28 day treatment period.
Arm/Group | Topicort® Topical Spray, 0.25%
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129
Other Adverse Events (participants affected / at risk) | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT02340169/Prot_SAP_000.pdf